CLINICAL TRIAL: NCT05612165
Title: Effectiveness and Safety of Transcranial Direct Current Stimulation for Pain Changes in Patients With Central Post-Stroke Pain
Brief Title: Effectiveness and Safety of tDCS for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-2022-001
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS group (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation(tDCS)
- Control group (Sham Comparator)
  Interventions: Device: Sham Transcranial Direct Current Stimulation(sham tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation(tDCS) — The tDCS intervention was conducted for 20 minutes(2000μA) each time, 5 times a week for 2 weeks, a total of 10 times.
  Arms: tDCS group
Device: Sham Transcranial Direct Current Stimulation(sham tDCS) — The sham tDCS intervention was conducted for 20 minutes(0μA) each time, 5 times a week for 2 weeks, a total of 10 times.
  Arms: Control group

SUMMARY:
The purpose of this study is to verify the effectiveness and safety of transcranial direct current stimulation in patients with central post-stroke pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 90 years old
2. Those who have been diagnosed with first-time stroke through doctors' clinical observation and brain imaging diagnosis
3. A person whose stroke lesions are cortex or subcortex
4. A person who satisfies 'Mandatory criteria'
5. Those with cognitive ability to understand and follow the researcher's instructions
6. Those who voluntarily agree to participate in this clinical trial and signed the agreement

Exclusion Criteria:

1. Those who have a fracture or have undergone orthopedic surgery
2. In case of accompanying serious neurological diseases
3. In case of major psychiatric diseases such as major depression disorders, schizophrenia, bipolar disorders, and dementia
4. Those with complex part pain syndrome by Budapest Criteria
5. If there is a cause of other pain in the relevant area, such as peripheral nerve damage
6. Persons included in the exclusion of transcranial direct current stimulation
7. If the researcher is judged to be judged that the participation in this study is not appropriate

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change of pain score in Brief Pain Inventory(BPI) | Baseline, after 2 weeks(after the end of intervention)
  Brief Pain Inventory(BPI) is used for measurement. The Brief Pain Inventory (BPI) is a tool used to assess pain severity and its impact on daily functions. The BPI typically uses an 11-point numeric rating scale (NRS) for its pain severity and pain interference items. Each item is rated from 0 to 10.
  Pain Severity: 0 (no pain) to 10 (pain as bad as you can imagine). Pain Interference: 0 (does not interfere) to 10 (completely interferes).

SECONDARY OUTCOMES:
Change of pain score in Neuropathic Pain Scale(NPS) | Baseline, after 2 weeks(after the end of intervention)
  Neuropathic Pain Scale(NPS) is used for measurement. The Neuropathic Pain Scale (NPS) is a tool used to assess the various qualities and intensities of neuropathic pain. Each Item: 0 (no pain or absence of the described pain quality) to 10 (the most intense pain or presence of the described pain quality imaginable).
Change of depression score in Beck Depression Inventory-II(BDI-II) | Baseline, after 2 weeks(after the end of intervention)
  Beck Depression Inventory-II(BDI-II) is used for measurement. The Beck Depression Inventory-II (BDI-II) is a widely used instrument for measuring the severity of depression. Minimum and Maximum Values: The BDI-II consists of 21 items, each rated on a 4-point scale ranging from 0 to 3. Total Score Range: 0 to 63. Each Item: 0 (symptom is absent) to 3 (severe level of the symptom).
Change of quality of life score in the EuroQol Five-dimensions-Three-Level Quality of Life Instrument(EQ-5D-3L) | Baseline, after 2 weeks(after the end of intervention)
  The EuroQol Five-dimensions-Three-Level Quality of Life Instrument(EQ-5D-3L) is used for measurement. The EuroQol Five-Dimensions-Three-Level Quality of Life Instrument (EQ-5D-3L) is a standardized instrument used to measure health-related quality of life. This utility score reflects the overall quality of life associated with each health state and typically ranges from -0.594 to 1 in the UK: A value closer to 1 indicates a better health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea